CLINICAL TRIAL: NCT02673684
Title: Double Blind, Randomized, Sham-Controlled Study on the Effects of Neuro-Stim System on Pain, Sleep, and Opioid Use in Pain Patients
Brief Title: Effects of Neuro-Stim System on Pain, Sleep, and Opioid Use
Acronym: NSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost funding from sponsor
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Collaborators: Innovative Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 390805
Record Dates: First submitted 2016-01-27; First posted 2016-02-04 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Pain (Visceral, Somatic, or Neuropathic)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Neurostim System (Sham NSS) (Sham Comparator): In this arm, the subject will receive the standard-of-care with regard to his pain management (which may or may not include opioids such as morphine). Additionally, the subject will receive a sham Neuro-Stim System device that will only be active for five minutes. Identical to the active device in placement, labeling, and packaging. It will remain on the subject's ear for 5 days at which point the subject may discard the device.
  Interventions: Device: Sham NSS
- Working Neurostim System (Working NSS) (Experimental): In this arm, the patient will receive the standard-of-care with regard to his pain management (which may or may not include opioids such as morphine). Additionally, the subject will receive an active Neuro-Stim System that generates electrical impulses that stimulate the neurovascular bundles in the ear. It will remain on subject's ear for 5 days at which point the subject may discard the device.
  Interventions: Device: Experimental NSS

INTERVENTIONS:
Device: Experimental NSS — 5-Day Active electro auricular device that delivers electrical impulses that stimulate the neurovascular bundles in the ear.
  Other Names: Electro Auricular Device
  Arms: Working Neurostim System (Working NSS)
Device: Sham NSS — (5 minute active) Electro Auricular Device that delivers electrical impulses to neurovascular bundles in the ear.
  Arms: Sham Neurostim System (Sham NSS)

SUMMARY:
The purpose of this study is to evaluate the ability of Neuro-Stim System, a non-pharmacologic alternative for pain management, to reduce pain and treat insomnia. Neuro-Stim System uses electrical current to stimulate neurovascular bundles (nerves) in the ear and possibly the autonomic nervous system.

DETAILED DESCRIPTION:
Pain is a complex problem that complicates recovery and rehabilitation after traumatic injury and surgery. The physician must balance pain management therapies against the potential for side effects and complications. Most of the treatment options for pain are pharmacological and have the potential for serious side effects and drug interactions. A non-pharmacological treatment would reduce the risk of adverse events and likely enhance the overall multimodal pain plan. The purpose of this study is to evaluate the effectiveness of Neuro-Stim System (NSS), a non-pharmacological option that uses electrical current to stimulate neurovascular bundles (nerves) in the ear and possibly the autonomic nervous system, to treat pain and improve sleep. Pain patients will be asked to participate in a study to evaluate the ability of Neuro-Stim System to reduce pain and to treat insomnia. NSS is a Federal Drug Administration (FDA) approved device intended to be used for chronic and acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be inpatients (at Walter Reed National Military Medical Center) at the time of study enrollment and study device placement.
* Any patient experiencing post-operative pain (visceral, somatic, or neuropathic) and has a pain score (measured via DVPRS v2.0) equal to or greater than 4 for at least 3 hours in the past 24 hours.
* Has an intact external ear where device can be placed
* The skin of the ear at placement site must be free of infection
* The participant cannot have been on regularly scheduled central acting opioids for more than 30 days continuously leading up to the initiation of the study. However, intermittent, breakthrough opioids are permissible, but the potential subject must have a current opioid prescription.
* The participant must have vital signs (HR/breathing/blood pressure) within normal limits.
* Able to understand English and verbalize their pain level.

Exclusion Criteria:

* Have inconsistent vital signs (fluctuating, extremely low blood pressure, tachycardia, etc.)
* Wear any time of implanted electrical device such as a brain shunt, vagal stimulator, pace maker, spinal pain pump, etc.
* Pregnant (by results of preoperative Human Chorionic Gonadotropin or hCG urine or blood testing)
* Has a history of skin allergy to metals
* unwilling to voluntarily participate
* hemophilia
* Psoriasis vulgaris on ears

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chester Buckenmaier, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham NSS: In this arm, the subject will receive the standard-of-care with regard to his pain management (which may or may not include opioids such as morphine). Additionally, the subject will receive a sham Neuro-Stim System device that will only be active for five minutes. Identical to the active device in placement, labeling, and packaging. It will remain on the subject's ear for 5 days at which point the subject may discard the device.
  Sham NSS: (5 minute active) Electro Auricular Device that delivers electrical impulses to neurovascular bundles in the ear.
- NSS (Working Device): In this arm, the patient will receive the standard-of-care with regard to his pain management (which may or may not include opioids such as morphine). Additionally, the subject will receive an active Neuro-Stim System that generates electrical impulses that stimulate the neurovascular bundles in the ear. It will remain on subject's ear for 5 days at which point the subject may discard the device.
  Experimental NSS: 5-Day Active electro auricular device that delivers electrical impulses that stimulate the neurovascular bundles in the ear.
Period: Overall Study
Arm/Group | Sham NSS | NSS (Working Device)
Started | 9 | 8
Completed | 0 | 0
Not Completed | 9 | 8
Not completed — Study not completed d/t loss of funding | 9 | 8

BASELINE CHARACTERISTICS:
Population: Study lost funding in the early stages therefore we were unable to collect enough data to do any analyzing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham NSS | NSS (Working Device) | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Measured Via the Defense and Veterans Pain Scale v2.0 (DVPRS)
Description: The primary outcome is pain measured by the Defense and Veterans Pain Rating Scale (DVPRS) from 0-10 at baseline, 15 minutes, and daily for 5 days after application.
  Rate the severity of your CURRENT pain:
  0 - No Pain
  1. - Hardly notice pain
  2. - Notice pain, does not interfere with activities
  3. - Sometimes distracts me
  4. - Distracts me, can do usual activities
  5. - Interrupts some activities
  6. - Hard to ignore, avoid usual activities
  7. - Focus of attention, prevents doing daily activities
  8. - Awful, hard to do anything
  9. - Can't bear pain, unable to do anything
  10. - As bad as it could be, nothing else matters
  Higher values represent worse outcomes
Time Frame: baseline to 5 days
Population: Sufficient data was not collected and the study was terminated. No data analysis was done due to loss of funding in the early stages of project.
Arm/Group | NSS (Working Device) | Sham NSS
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Modified PROMIS for Pain Intensity
Description: Use the scale to answer the following questions for Pain Intensity in the past 24 hours,
  1=had no pain 2=Mild 3= Moderate 4= Severe 5=Very Severe
  1. How intense was your pain at its worst?
  2. How intense was your average pain?
  3. What is your level of pain right now?
  Higher values represent worse outcomes
Time Frame: baseline to 10 days
Population: as for outcome 1
Arm/Group | Sham NSS | NSS (Working Device)
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Modified PROMIS for Pain Interference
Description: Use the following scale to to answer the questions about Pain Interference in the last 24 hours
  1=Not at all 2=A little bit 3= Somewhat 4= Quite a bit 5=Very much
  1. How much did pain interfere with your enjoyment of life?
  2. How much did pain interfere with your ability to concentrate?
  3. How much did pain interfere with your day to day activities?
Time Frame: baseline to 10 days
Population: No data analysis was done due to loss of funding in the early stages of project.
Arm/Group | NSS (Working Device) | Sham NSS
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Modified PROMIS for Sleep Disturbance
Description: Use the scale to answer the following question regarding Sleep Disturbance in the past 24 hours
  1=Very Poor 2=Poor 3= Fair 4= Good 5=Very Good
  1. My sleep quality was...
  Use the scale to answer the following questions regarding Sleep Disturbance in the past 24 hours
  1=Not at all 2=A little bit 3= Somewhat 4= Quite a bit 5=Very much
  1. My sleep was refreshing…
  2. I had a problem with my sleep…
  3. I had difficulty falling asleep…
Time Frame: baseline to 10 days
Population: No data analysis was done due to loss of funding in the early stages of project.
Arm/Group | NSS (Working Device) | Sham NSS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: STUDY LOST FUNDING IN THE EARLY STAGES The total duration of this study was 3 months, we did not have any adverse events to report.
Description: We did not have any adverse events to report for the duration of the study.
Arm/Group | Sham NSS | NSS (Working Device)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Lost funding in the early stages of the project which ended recruitment to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No